CLINICAL TRIAL: NCT00575549
Title: Prospective Analysis and Comparison of Conventional Stress Echocardiograms and Real-Time Myocardial Contrast Stress Echocardiogram; for Bristol-Myers Squibb Medical Imaging: The Definity RT-P During DSE Database
Brief Title: Prospective Analysis and Comparison of Stress Echo to Real-Time Myocardial Contrast Stress Echo
Status: No longer available | Type: Expanded Access
Sponsor: University of Nebraska (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 0311-07-FB
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Evaluation of Troponin I Levels
MeSH Terms: interventions — perflutren

INTERVENTIONS:
Other: Dobutamine: Perflutren Lipid Microsphere — Dobutamine with starting dose of 10 micrograms/kg/min and increased gradually to a maximum dose of 50 micrograms/kg/min Definity will be infused continuously at a rate of 4mL/min
  Other Names: Definity

SUMMARY:
The purpose of this study is to prospectively analyze and compare conventional stress echocardiograms and real-time myocardial contrast stress echocardiograms; and to determine the effect of contrast agents used during real-time myocardial contrast stress echocardiograms on serum troponin I levels.

DETAILED DESCRIPTION:
To compare two different stress echocardiograms (conventional Stress echocardiograms or Real-time Myocardial Contrast Stress Echocardiograms) that are in routine clinical use. The information, including the digital images that are collected during the stress tests is used to determine if the usse of specialized imaging techniques and ultrasound contrast can better detect blockage in blood flow to the heart and predict how patients outcome may be affected by this detection of a blockage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age > 19 years
* Scheduled for a stress echocardiography
* Are conscious and coherent, and able to communicate effectively with trial personnel
* For troponin evaluation, only hospitalized patients who had a troponin level drawn in the morning of and prior to stress echocardiogram will be included.

Exclusion Criteria:

* Pregnant and breast feeding women are excluded from participation because of the possibility of a bias as CSE is routinely used in pregnant patients secondary to lack of human studies to determine the fetal risk of use of Definity.
* Age < 19 years old
* Known or suspected hypersensitivity to ultrasound contrast agents or other drugs used for the study
* Possibility that potential subject may be pregnant
* Studies where RT-MCE was specifically requested by the ordering physician

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States